CLINICAL TRIAL: NCT03833778
Title: Kids + Adolescents Research Learning On Tablet Teaching Aachen
Acronym: KARLOTTA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: RWTH Aachen University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 18-007
Record Dates: First submitted 2019-02-06; First posted 2019-02-07 (Actual); Last update posted 2022-10-26 (Actual); Status verified 2022-10

CONDITIONS: Chronic Inflammatory Intestinal Diseases (CED)

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Other): Answering disease related questions during playing a tablet game
  Interventions: Other: intervention group
- control group (No Intervention)

INTERVENTIONS:
Other: intervention group — The CED patients play the tablet-CED-quiz, while they wait for their doctor's appointment, so that gaps in the CED knowledge can be clarified during the doctor's consultation.
  Arms: Intervention group

SUMMARY:
The aim of this study plan is to implement a tablet quiz in the German-speaking area, in order to test the specific knowledge about chronic inflammatory intestinal diseases (CED) concerning pediatric patients in the context of an age-appropriated and interesting digital playing environment, and to process knowledge gaps at the subsequent doctor's contact. The quiz should be combined with a game and can be performed by the patients, while they wait in the ambulance for their doctor's appointment. The investigator's goals are to grasp playfully gaps in the CED knowledge regarding the patients and to use these in the following consulting hour for clarification and advice in line with a better understanding of the disease. With this, the specific knowledge, the understanding of the disease, the therapeutic adherence, and the self-efficacy should improve the self-responsible handling of the disease. In particular, the willingness of the group of older teenagers to transit into the adult medicine can be collected and processed. The investigators want to check the efficacy in a randomized, controlled study with two groups of 15 pediatric CED patients. The hypothesis is that the additional play of the tablet-CED-quiz and the individualized advice have a positive impact on the CED knowledge, the disease activity, the CED-related life quality and the willingness of teenagers for transition.

ELIGIBILITY:
Inclusion Criteria:

* Female and male children and young adults between 8-21 years
* Diagnosis Morbus Crohn, Colitis ulcerosa or Colitis indeterminate
* Clarification and signed Informed Consent Form
* Patients must know how to write and read in German
* Patients must be able to play independently on the tablet

Exclusion Criteria:

* Age < 8 years or > 21 years
* Illiteracy
* Mental or psychomotor disability

Ages: 8 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30 (Actual)
Dates: Start 2019-02-05 (Actual); Primary Completion 2020-07-30 (Actual); Study Completion 2020-07-31 (Actual)

PRIMARY OUTCOMES:
knowledge test | 12 months
  Comparing point values of the baseline tablet quiz and final test regarding the CED knowledge

CONTACTS AND LOCATIONS:
Overall Officials: Angeliki Pappa, Dr. med., Principal Investigator — Clinic for Pediatrics and Youth Medicine, University Hospital of RWTH Aachen University
Locations (1):
- Clinic for Pediatrics and Youth Medicine, University Hospital of RWTH Aachen University, Aachen, North Rhine-Westphalia, Germany

IPD SHARING:
Plan to Share IPD: No